CLINICAL TRIAL: NCT02508649
Title: A Double-blind, Randomised, Placebo-Controlled, Phase 2b/3 Adaptive Clinical Trial Investigating the Efficacy and Safety of Selepressin as Treatment for Patients With Vasopressor-dependent Septic Shock
Brief Title: Selepressin Evaluation Programme for Sepsis-Induced Shock - Adaptive Clinical Trial
Acronym: SEPSIS-ACT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to futility
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000133; 2014-003973-41 (EudraCT Number)
Record Dates: First submitted 2015-07-17; First posted 2015-07-27 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-09

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Selepressin 1 (Experimental): Starting dose 1.7 ng/kg/min
  Interventions: Drug: selepressin
- Selepressin 2 (Experimental): Starting dose 2.5 ng/kg/min
  Interventions: Drug: selepressin
- Selepressin 3 (Experimental): Starting dose 3.5 ng/kg/min
  Interventions: Drug: selepressin
- Selepressin 4 (Experimental): Starting dose 5.0 ng/kg/min
  The highest dosing regimen of selepressin was not investigated in the trial as the desired primary outcome for selepressin 3 arm was not achieved, and the trial was terminated for futility.
  Interventions: Drug: selepressin

INTERVENTIONS:
Drug: selepressin
  Arms: Selepressin 1; Selepressin 2; Selepressin 3; Selepressin 4
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomised, placebo-controlled, two-part adaptive clinical trial. The trial is designed to investigate the efficacy and safety of multiple dosing regimens of selepressin and to confirm the efficacy and safety of one dosing regimen in treatment of adult patients with septic shock requiring vasopressor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Proven or suspected infection
* Septic shock defined as hypotension requiring vasopressor treatment despite adequate fluid resuscitation
* Informed consent obtained in accordance with local regulations

Exclusion Criteria:

* Not possible to initiate trial drug treatment within 12 hours from onset of vasopressor treatment for septic shock
* Primary cause of hypotension not due to sepsis
* Previous severe sepsis with intensive care unit admission within this hospital stay
* Known/suspected acute mesenteric ischaemia
* Suspicion of concomitant acute coronary syndrome based on clinical symptoms and/or ECG during this episode of septic shock
* Chronic mechanical ventilation for any reason OR severe chronic obstructive pulmonary disease (COPD) requiring either continuous daily oxygen use during the preceding 30 days or mechanical ventilation (for acute exacerbation of COPD) during the preceding 30 days
* Received bone marrow transplant during the preceding 6 months or chemotherapy during the preceding 30 days for lymphoma or leukemia
* Known to be pregnant
* Decision to limit full care taken before obtaining informed consent
* Use of vasopressin in the past 12 hours prior to start of trial drug treatment or use of terlipressin within 7 days prior to start of trial drug treatment
* Prior enrolment in the trial
* Prior use of an investigational medicinal product within the last month OR planned or concurrent participation in a clinical trial for any investigational drug or investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (21):
- United States (17):
  - Memorial Hospital, Colorado Springs, Colorado
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Healthsystem Research Institute, Evanston, Illinois
  - Stormont Vail Health Care, Topeka, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - HealthPartners Speciality Clinics, Saint Paul, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - St Vincent Mercy Medical Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Cliniques Universitaires Saint-Luc (there may be other sites in this country), Brussels, Belgium
- Aalborg Universitetshospital (there may be other sites in this country), Aalborg, Denmark
- Centre Hospitalier et Universitaire de Limoges (there may be other sites in this country), Limoges, France
- Radboud University Nijmegen Medical Centre (there may be other sites in this country), Nijmegen, Netherlands

REFERENCES:
- [Derived] Laterre PF, Berry SM, Blemings A, Carlsen JE, Francois B, Graves T, Jacobsen K, Lewis RJ, Opal SM, Perner A, Pickkers P, Russell JA, Windelov NA, Yealy DM, Asfar P, Bestle MH, Muller G, Bruel C, Brule N, Decruyenaere J, Dive AM, Dugernier T, Krell K, Lefrant JY, Megarbane B, Mercier E, Mira JP, Quenot JP, Rasmussen BS, Thorsen-Meyer HC, Vander Laenen M, Vang ML, Vignon P, Vinatier I, Wichmann S, Wittebole X, Kjolbye AL, Angus DC; SEPSIS-ACT Investigators. Effect of Selepressin vs Placebo on Ventilator- and Vasopressor-Free Days in Patients With Septic Shock: The SEPSIS-ACT Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1476-1485. doi: 10.1001/jama.2019.14607. PMID 31577035
- [Derived] Lewis RJ, Angus DC, Laterre PF, Kjolbye AL, van der Meulen E, Blemings A, Graves T, Russell JA, Carlsen JE, Jacobsen K, Yealy DM, Opal SM, Windelov NA, Francois B, Perner A, Pickkers P, Berry SM. Rationale and Design of an Adaptive Phase 2b/3 Clinical Trial of Selepressin for Adults in Septic Shock. Selepressin Evaluation Programme for Sepsis-induced Shock-Adaptive Clinical Trial. Ann Am Thorac Soc. 2018 Feb;15(2):250-257. doi: 10.1513/AnnalsATS.201708-669SD. PMID 29388815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 sites were authorized to recruit subjects for the trial between July 2015 and August 2017. Eleven of these sites did not recruit any subjects. The trial sites that randomized subjects to the trial were: 11 in Belgium, 5 in Denmark, 17 in France, 5 in the Netherlands, and 14 in the United States of America (USA).
Pre-assignment Details: A total of 6377 subjects were screened, of which 868 subjects were randomized (585 subjects were allocated to selepressin [three doses] and 283 subjects were allocated to placebo).
  Up to four dosing regimens of selepressin were planned to be investigated in the trial. However, the highest dosing regimen was not used.
Groups:
- Placebo: Sterile 0.9% sodium chloride solution given as an infusion, was used as the placebo.
- Selepressin 2.5 ng/kg/Min: Starting dose: 1.7 ng/kg/min selepressin; Maximum dose: 2.5 ng/kg/min selepressin, given as an infusion.
- Selepressin 3.75 ng/kg/Min: Starting dose: 2.5 ng/kg/min selepressin; Maximum dose: 3.75 ng/kg/min selepressin, given as an infusion.
- Selepressin 5.25 ng/kg/Min: Starting dose: 3.5 ng/kg/min selepressin; Maximum dose: 5.25 ng/kg/min selepressin, given as an infusion.
Period: Overall Study
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min
Started | 283 | 197 | 189 | 199
Dosed | 266 | 191 | 177 | 194
Completed | 265 | 184 | 174 | 189
Not Completed | 18 | 13 | 15 | 10
Not completed — Withdrawal by Subject | 4 | 6 | 5 | 6
Not completed — Investigator withdrew the subject | 1 | 2 | 1 | 0
Not completed — Post randomization screening failure | 12 | 4 | 9 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised of all the subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Total
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 828
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (14.56) | 66.0 (12.76) | 67.2 (13.13) | 66.8 (12.47) | 66.3 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 80 | 70 | 70 | 341
  Male | 145 | 111 | 107 | 124 | 487
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 1 | 4 | 12
  Not Hispanic or Latino | 262 | 188 | 176 | 190 | 816
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 5 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 11 | 7 | 25
  White | 260 | 186 | 161 | 183 | 790
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Number analyzed differs from the overall population as baseline body mass index (BMI) was not calculated for some of the subjects. The reason is that data was not collected for all subjects.
  kg/m^2
    number analyzed (Participants) | 265 | 191 | 176 | 192 | 824
    (all) | 27.47 (7.234) | 27.56 (8.778) | 28.04 (7.885) | 27.98 (8.565) | 27.73 (8.055)

OUTCOME MEASURES:

1. Primary Outcome: Vasopressor- and Mechanical Ventilator-free Days (PVFDs)
Description: Composite endpoint defined as number of days from start of treatment to 30 days thereafter during which subject is:
  1. Alive. However, if patient dies within these 30-days then PVFDs will be zero even if there is a period during which subject is alive and free of both vasopressor treatment and mechanical ventilation;
  2. Free of treatment with vasopressors: Less than 60 min during any contiguous 24-h period. If a patient requires vasopressors longer than 60 min in total during any 24-h period, the intervening intervals during which they are free of vasopressors will not be included in the determination of PVFDs;
  3. Free of any mechanical ventilation: Less than 60 min during any contiguous 24-h period. If a patient requires mechanical ventilation longer than 60 min in total during any 24-h period, the intervening intervals during which they are not receiving mechanical ventilation will not be included in the period free of mechanical ventilation in the determination of PVFDs.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed. The primary comparison to determine statistical and clinical significance was between all subjects in all selepressin arms (pooled together and treated as a single arm) and all subjects in the placebo arm, to control Type 1 error.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Groups:
- Selepressin Pooled: All selepressin arms pooled together and treated as a single arm.
Arm/Group | Placebo | Selepressin Pooled
Number analyzed (Participants) | 266 | 562
days | 14.45 [12.82 to 16.09] | 15.00 [13.77 to 16.23]
Statistical Analysis 1: Comparison: Placebo vs Selepressin Pooled; The primary endpoint was analyzed using a van Elteren test. The analysis included a test of superiority using a two-sided 5% significance level; Test type: Superiority; p = 0.3015, van Elteren test; Treatment difference = 0.55, 95% CI 2-sided [-1.34 to 2.43]

2. Secondary Outcome: All-cause Mortality
Description: All-cause mortality defined as the percentage of subjects that have died, regardless of cause.
Time Frame: At Day 90
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Selepressin Pooled
Number analyzed (Participants) | 257 | 526
percentage of subjects | 39.44 | 40.59
Statistical Analysis 1: Comparison: Placebo vs Selepressin Pooled; Mortality was analyzed using a logistic regression model with the individual sequential organ failure assessment (SOFA) scores and age as covariates and treatment arm as factor; Test type: Superiority; p = 0.7694, Regression, Logistic; Odds Ratio (OR) = 1.049, 95% CI 2-sided [0.762 to 1.445] — An odds ratio < 1 in proportion of subjects dying indicates lower mortality in the selepressin group

3. Secondary Outcome: Renal Replacement Therapy (RRT)-Free Days
Description: RRT-free days was defined as the number of days a subject is free of treatment with any form of RRT (continuous RRT, intermittent hemodialysis or peritoneal dialysis) and the intermittent periods were not included.
  RRT-free days was analyzed excluding subjects on RRT for chronic renal failure at time of randomization.
Time Frame: Up to Day 30
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Selepressin Pooled
Number analyzed (Participants) | 261 | 550
days | 18.21 [16.14 to 20.29] | 18.50 [17.03 to 19.98]
Statistical Analysis 1: Comparison: Placebo vs Selepressin Pooled; This endpoint was analyzed using a van Elteren test. The analysis was a test of superiority using a two-sided 5% significance level; Test type: Superiority; p = 0.8458, van Elteren test; Treatment difference = 0.29, 95% CI 2-sided [-2.07 to 2.65]

4. Secondary Outcome: Intensive Care Unit (ICU)-Free Days
Description: The ICU free days, as for the PVFDs, reflect the time from last discharge of the ICU to Day 30 with an absolute penalty for mortality, i.e., any subject that died within this 30-day period was assigned zero value).
Time Frame: Up to Day 30
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Selepressin Pooled
Number analyzed (Participants) | 266 | 562
days | 12.15 [10.66 to 13.64] | 12.64 [11.51 to 13.76]
Statistical Analysis 1: Comparison: Placebo vs Selepressin Pooled; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4124, van Elteren test; Treatment difference = 0.49, 95% CI 2-sided [-1.22 to 2.19]

5. Secondary Outcome: Vasopressor-free Days up to Day 30
Description: Number of days from start of treatment to 30 days thereafter during which the subject is free of treatment with vasopressors, i.e. less than 60 min during any contiguous 24-h period.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
days | 25.30 [0.00 to 28.30] | 25.60 [0.00 to 28.60] | 23.30 [0.00 to 28.60] | 25.30 [0.00 to 28.80] | 25.10 [0.00 to 28.70]

6. Secondary Outcome: Mechanical Ventilator-free Days up to Day 30
Description: Number of days from start of treatment to 30 days thereafter during which the subject is free of any mechanical ventilation, i.e. less than 60 min during any contiguous 24-h period.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
days | 19.80 [0.00 to 29.40] | 18.90 [0.00 to 30.00] | 17.20 [0.00 to 29.10] | 17.50 [0.00 to 29.50] | 17.50 [0.00 to 29.80]

7. Secondary Outcome: Duration of Septic Shock (i.e. Vasopressor Use) up to Day 30
Description: The duration of septic shock was defined as the cumulative periods (>1 h), from start of investigational medicinal product (IMP) treatment until Day 30, on IMP or vasopressors.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
days | 2.220 [1.110 to 4.420] | 1.660 [0.800 to 2.990] | 1.790 [0.810 to 4.370] | 1.465 [0.750 to 3.530] | 1.635 [0.770 to 3.650]

8. Secondary Outcome: Duration of Mechanical Ventilation up to Day 30
Description: The duration of mechanical ventilation was defined as the cumulative periods (>1 h), from start of the IMP treatment until Day 30, on mechanical ventilation.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
days | 2.255 [0.000 to 8.710] | 1.690 [0.000 to 8.250] | 2.800 [0.100 to 8.880] | 1.910 [0.000 to 7.680] | 1.990 [0.000 to 8.250]

9. Secondary Outcome: The Percentage of Subjects With RRT up to Day 30 (Counting Subjects Who Died as on RRT and Excluding Subjects on RRT for Chronic Renal Failure at the Time of Randomization)
Description: Renal replacement therapy is defined as continuous RRT, intermittent hemodialysis, or peritoneal dialysis. In order to ensure that any reduction in the incidence of RRT was not caused by an increase in mortality, all subjects dying within the 30-day period were counted as on RRT.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 261 | 187 | 174 | 189 | 550
Participants
  No | 135 | 102 | 89 | 100 | 291
  Yes | 126 | 85 | 85 | 89 | 259

10. Secondary Outcome: Duration of RRT up to Day 90 (Excluding Subjects on RRT for Chronic Failure at the Time of Randomization)
Description: The duration of RRT was defined as the cumulative periods (>1 h) from start of IMP until Day 90 with RRT (continuous renal replacement therapy, intermittent hemodialysis, or peritoneal dialysis).
  Subjects on RRT for chronic renal failure at time of randomization were not included in the analysis.
Time Frame: Up to Day 90
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 261 | 187 | 174 | 189 | 550
days | 1.634 (5.5380) | 1.739 (5.5593) | 1.876 (6.0300) | 2.459 (10.1365) | 2.030 (7.5640)

11. Secondary Outcome: Overall and Individual Organ (Cardiovascular, Respiratory, Renal, Hepatic, Coagulation) Scores Using a Modified Version of the SOFA up to Day 7 or Until ICU Discharge
Description: The presence of 5 organ dysfunctions (cardiovascular, respiratory, renal, hepatic, coagulation) was assessed using a modified Sequential Organ Failure Assessment (SOFA) (i.e. SOFA except the Glasgow Coma Scale). In addition, any dose of vasopressors or positive ionotropes will attribute 3 or 2 points on the cardiovascular scale, respectively.
  Each organ has a possible dysfunction score of 0 (no organ dysfunction) to 4 (dysfunctional organ), for a total modified SOFA score range of 0 (no organ dysfunction) to 23 (all organs with dysfunction).
Time Frame: Days 1, 3, and 7 or discharge from ICU
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Selepressin Pooled
Number analyzed (Participants) | 263 | 555
score on a scale
  Overall score (Day 1): number analyzed (Participants) | 247 | 515
  Overall score (Day 1) | 9.95 [9.31 to 10.60] | 9.44 [9.00 to 9.89]
  Overall score (Day 3): number analyzed (Participants) | 240 | 474
  Overall score (Day 3) | 8.95 [8.30 to 9.59] | 9.06 [8.60 to 9.51]
  Overall score (Day 7): number analyzed (Participants) | 182 | 382
  Overall score (Day 7) | 8.08 [7.41 to 8.76] | 8.63 [8.17 to 9.10]
  Individual (Respiratory) score Day 1: number analyzed (Participants) | 256 | 532
  Individual (Respiratory) score Day 1 | 2.58 [2.45 to 2.71] | 2.50 [2.41 to 2.59]
  Individual (Respiratory) score Day 3: number analyzed (Participants) | 245 | 483
  Individual (Respiratory) score Day 3 | 2.43 [2.30 to 2.56] | 2.40 [2.31 to 2.49]
  Individual (Respiratory) score Day 7: number analyzed (Participants) | 186 | 388
  Individual (Respiratory) score Day 7 | 2.38 [2.24 to 2.52] | 2.41 [2.31 to 2.50]
  Individual (Cardiovascular) score Day 1 | 3.66 [3.47 to 3.85] | 3.23 [3.10 to 3.36]
  Individual (Cardiovascular) score Day 3: number analyzed (Participants) | 250 | 496
  Individual (Cardiovascular) score Day 3 | 2.33 [2.14 to 2.53] | 2.08 [1.95 to 2.22]
  Individual (Cardiovascular) score Day 7: number analyzed (Participants) | 188 | 396
  Individual (Cardiovascular) score Day 7 | 1.79 [1.58 to 1.99] | 1.65 [1.51 to 1.79]
  Individual (Renal) score Day 1 | 1.64 [1.47 to 1.81] | 1.59 [1.48 to 1.71]
  Individual (Renal) score Day 3: number analyzed (Participants) | 250 | 496
  Individual (Renal) score Day 3 | 1.52 [1.35 to 1.69] | 1.61 [1.49 to 1.73]
  Individual (Renal) score Day 7: number analyzed (Participants) | 188 | 396
  Individual (Renal) score Day 7 | 1.46 [1.28 to 1.64] | 1.63 [1.50 to 1.75]
  Individual (Coagulation) score Day 1: number analyzed (Participants) | 260 | 551
  Individual (Coagulation) score Day 1 | 1.15 [1.00 to 1.30] | 1.27 [1.16 to 1.37]
  Individual (Coagulation) score Day 3: number analyzed (Participants) | 248 | 495
  Individual (Coagulation) score Day 3 | 1.50 [1.35 to 1.66] | 1.73 [1.62 to 1.84]
  Individual (Coagulation) score Day 7: number analyzed (Participants) | 187 | 395
  Individual (Coagulation) score Day 7 | 1.30 [1.14 to 1.46] | 1.53 [1.42 to 1.64]
  Individual (Liver) score Day 1: number analyzed (Participants) | 256 | 540
  Individual (Liver) score Day 1 | 0.87 [0.71 to 1.03] | 0.72 [0.61 to 0.83]
  Individual (Liver) score Day 3: number analyzed (Participants) | 247 | 488
  Individual (Liver) score Day 3 | 1.11 [0.95 to 1.28] | 1.07 [0.95 to 1.18]
  Individual (Liver) score Day 7: number analyzed (Participants) | 185 | 391
  Individual (Liver) score Day 7 | 1.17 [1.00 to 1.35] | 1.35 [1.23 to 1.46]
Statistical Analysis 1: Comparison: Placebo vs Selepressin Pooled; Overall score using a modified version of the SOFA on Day 1; Test type: Other; p = 0.2009, ANCOVA; Treatment difference = -0.51, 95% CI 2-sided [-1.30 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs Selepressin Pooled; Overall score using a modified version of the SOFA on Day 3; Test type: Other; p = 0.7894, ANCOVA; Treatment difference = 0.11, 95% CI 2-sided [-0.68 to 0.90]
Statistical Analysis 3: Comparison: Placebo vs Selepressin Pooled; Overall score using a modified version of the SOFA on Day 7; Test type: Other; p = 0.1888, ANCOVA; Treatment difference = 0.55, 95% CI 2-sided [-0.27 to 1.37]
Statistical Analysis 4: Comparison: Placebo vs Selepressin Pooled; Individual organ (respiratory) score using a modified version of the SOFA on Day 1; Test type: Other; p = 0.2997, ANCOVA; Treatment difference = -0.08, 95% CI 2-sided [-0.24 to 0.07]
Statistical Analysis 5: Comparison: Placebo vs Selepressin Pooled; Individual organ (respiratory) score using a modified version of the SOFA on Day 3; Test type: Other; p = 0.6796, ANCOVA; Treatment difference = -0.03, 95% CI 2-sided [-0.19 to 0.12]
Statistical Analysis 6: Comparison: Placebo vs Selepressin Pooled; Individual organ (respiratory) score using a modified version of the SOFA on Day 7; Test type: Other; p = 0.7467, ANCOVA; Treatment difference = 0.03, 95% CI 2-sided [-0.14 to 0.19]
Statistical Analysis 7: Comparison: Placebo vs Selepressin Pooled; Individual organ (cardiovascular) score using a modified version of the SOFA on Day 1; Test type: Other; p = 0.0003, ANCOVA; Treatment difference = -0.42, 95% CI 2-sided [-0.65 to -0.19]
Statistical Analysis 8: Comparison: Placebo vs Selepressin Pooled; Individual organ (cardiovascular) score using a modified version of the SOFA on Day 3; Test type: Other; p = 0.0349, ANCOVA; Treatment difference = -0.25, 95% CI 2-sided [-0.49 to -0.02]
Statistical Analysis 9: Comparison: Placebo vs Selepressin Pooled; Individual organ (cardiovascular) score using a modified version of the SOFA on Day 7; Test type: Other; p = 0.2787, ANCOVA; Treatment difference = -0.14, 95% CI 2-sided [-0.39 to 0.11]
Statistical Analysis 10: Comparison: Placebo vs Selepressin Pooled; Individual organ (renal) score using a modified version of the SOFA on Day 1; Test type: Other; p = 0.6476, ANCOVA; Treatment difference = -0.05, 95% CI 2-sided [-0.26 to 0.16]
Statistical Analysis 11: Comparison: Placebo vs Selepressin Pooled; Individual organ (renal) score using a modified version of the SOFA on Day 3; Test type: Other; p = 0.4313, ANCOVA; Treatment difference = 0.08, 95% CI 2-sided [-0.13 to 0.29]
Statistical Analysis 12: Comparison: Placebo vs Selepressin Pooled; Individual organ (renal) score using a modified version of the SOFA on Day 7; Test type: Other; p = 0.1334, ANCOVA; Treatment difference = 0.17, 95% CI 2-sided [-0.05 to 0.39]
Statistical Analysis 13: Comparison: Placebo vs Selepressin Pooled; Individual organ (coagulation) score using a modified version of the SOFA on Day 1; Test type: Other; p = 0.2126, ANCOVA; Treatment difference = 0.12, 95% CI 2-sided [-0.07 to 0.30]
Statistical Analysis 14: Comparison: Placebo vs Selepressin Pooled; Individual organ (coagulation) score using a modified version of the SOFA on Day 3; Test type: Other; p = 0.0174, ANCOVA; Treatment Difference = 0.23, 95% CI 2-sided [0.04 to 0.41]
Statistical Analysis 15: Comparison: Placebo vs Selepressin Pooled; Individual organ (coagulation) score using a modified version of the SOFA on Day 7; Test type: Other; p = 0.0194, ANCOVA; Treatment difference = 0.23, 95% CI 2-sided [0.04 to 0.43]
Statistical Analysis 16: Comparison: Placebo vs Selepressin Pooled; Individual organ (liver) score using a modified version of the SOFA on Day 1; Test type: Other; p = 0.1284, ANCOVA; Treatment difference = -0.15, 95% CI 2-sided [-0.35 to 0.04]
Statistical Analysis 17: Comparison: Placebo vs Selepressin Pooled; Individual organ (liver) score using a modified version of the SOFA on Day 3; Test type: Other; p = 0.6542, ANCOVA; Treatment difference = -0.05, 95% CI 2-sided [-0.25 to 0.15]
Statistical Analysis 18: Comparison: Placebo vs Selepressin Pooled; Individual organ (liver) score using a modified version of the SOFA on Day 7; Test type: Other; p = 0.1079, ANCOVA; Treatment difference = 0.17, 95% CI 2-sided [-0.04 to 0.38]

12. Secondary Outcome: Percentage of Subjects With New Organ Dysfunction and New Organ Failure (Based on the SOFA Score) up to Day 7 and Day 30
Description: The presence of 5 organ dysfunctions (cardiovascular, respiratory, renal, hepatic, coagulation) was assessed using a SOFA score. Each organ has a possible dysfunction score of 0 (no organ dysfunction) to 4 (all organs with dysfunction).
  Incidence of new organ dysfunction is defined as an increase ≥ 1 from baseline to post baseline up until the end of the period (e.g. going from 1-2) in any of the individual SOFA scores.
  Incidence of new organ failures is defined as a change in any of the individual SOFA scores from (0-2) at baseline to (3-4) post baseline up until the end of the period (Day 7 or 30) (if the SOFA scores goes from (0-2) to (3-4) and back to (0-2) again within the period, that will still count as a new organ failure).
  Percentage of subjects with new organ dysfunction and new organ failure (based on the SOFA Score) up to Day 7 and Day 30 are reported.
Time Frame: Up to Day 7 and Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Placebo | Selepressin Pooled
Number analyzed (Participants) | 256 | 536
percentage of subjects
  New organ dysfunction (Day 7) | 76.41 [70.42 to 81.51] | 81.95 [77.92 to 85.38]
  New organ dysfunction (Day 30) | 80.44 [74.80 to 85.07] | 84.08 [80.21 to 87.31]
  New organ failure (Day 7) | 44.18 [37.67 to 50.90] | 47.39 [42.70 to 52.12]
  New organ failure (Day 30) | 56.91 [50.23 to 63.35] | 57.15 [52.39 to 61.78]
Statistical Analysis 1: Comparison: Placebo vs Selepressin Pooled; Percentage of subjects with new organ dysfunction up to Day 7; Test type: Other; p = 0.0630, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.98 to 2.00] — Odds ratio is equal to Selepressin pooled/Placebo
Statistical Analysis 2: Comparison: Placebo vs Selepressin Pooled; Percentage of subjects with new organ dysfunction up to Day 30; Test type: Other; p = 0.1875, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.89 to 1.86] — Odds ratio is equal to Selepressin pooled/Placebo
Statistical Analysis 3: Comparison: Placebo vs Selepressin Pooled; Percentage of subjects with new organ failure up to Day 7; Test type: Other; p = 0.4382, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.82 to 1.58] — Odds ratio is equal to Selepressin pooled/Placebo
Statistical Analysis 4: Comparison: Placebo vs Selepressin Pooled; Percentage of subjects with new organ failure up to Day 30; Test type: Other; p = 0.9529, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.73 to 1.39] — Odds ratio is equal to Selepressin pooled/Placebo

13. Secondary Outcome: ICU Length of Stay up to Day 30
Description: ICU length of stay is defined as the cumulative periods (>1 h) spent in ICU from start of IMP to 30 days after.
Time Frame: Up to Day 30
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
days | 6.755 [3.110 to 16.110] | 4.940 [2.500 to 13.530] | 6.460 [2.880 to 15.530] | 5.960 [2.790 to 14.380] | 5.695 [2.710 to 14.430]

14. Secondary Outcome: All-cause Mortality (Defined as the Percentage of Subjects That Have Died, Regardless of Cause) at Day 30 and Day 180
Description: All-cause mortality defined as the percentage of subjects that have died, regardless of cause.
Time Frame: At Day 30 and Day 180
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
Participants
  Day 30: number analyzed (Participants) | 265 | 187 | 176 | 189 | 552
  Day 30: No | 174 | 121 | 114 | 124 | 359
  Day 30: Yes | 91 | 66 | 62 | 65 | 193
  Day 180: number analyzed (Participants) | 263 | 184 | 172 | 187 | 543
  Day 180: No | 147 | 104 | 96 | 102 | 302
  Day 180: Yes | 116 | 80 | 76 | 85 | 241

15. Secondary Outcome: Daily Fluid Balance Until ICU Discharge (for a Maximum of 7 Days)
Description: Fluid balance (as a rate of time) calculated for fluid administered during episode of severe sepsis/septic shock will be presented until ICU discharge (for a maximum of 7 days).
Time Frame: Baseline and Days 1-7
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
mL/h
  Baseline: number analyzed (Participants) | 265 | 187 | 177 | 194 | 558
  Baseline | 339.10 (236.53) | 342.23 (218.17) | 365.14 (255.92) | 350.51 (278.28) | 352.38 (252.01)
  Day 1: number analyzed (Participants) | 265 | 191 | 177 | 194 | 562
  Day 1 | 104.74 (110.40) | 95.14 (116.90) | 86.80 (111.86) | 66.68 (96.94) | 82.68 (109.24)
  Day 2: number analyzed (Participants) | 241 | 175 | 160 | 181 | 516
  Day 2 | 51.78 (79.27) | 52.75 (74.12) | 48.95 (65.47) | 44.35 (73.82) | 48.62 (71.39)
  Day 3: number analyzed (Participants) | 214 | 148 | 147 | 157 | 452
  Day 3 | 19.71 (79.94) | 24.87 (65.20) | 33.34 (67.61) | 29.14 (75.19) | 29.11 (69.52)
  Day 4: number analyzed (Participants) | 201 | 130 | 130 | 139 | 399
  Day 4 | 2.34 (75.41) | 6.76 (59.14) | 22.28 (70.95) | 19.50 (66.09) | 16.25 (65.76)
  Day 5: number analyzed (Participants) | 173 | 105 | 114 | 124 | 343
  Day 5 | -0.30 (72.84) | 1.08 (62.02) | 5.94 (71.72) | 3.06 (62.49) | 3.41 (65.40)
  Day 6: number analyzed (Participants) | 154 | 88 | 92 | 109 | 289
  Day 6 | -4.70 (61.16) | -12.19 (80.30) | -3.49 (75.52) | -5.91 (64.72) | -7.05 (73.03)
  Day 7: number analyzed (Participants) | 139 | 84 | 87 | 97 | 268
  Day 7 | -5.84 (62.52) | -7.36 (63.51) | 4.17 (67.38) | -12.71 (58.19) | -5.55 (63.12)

16. Secondary Outcome: Cumulative Fluid Balance Until ICU Discharge (for a Maximum of 7 Days)
Description: Cumulative fluid balance (total volume) calculated for fluid administered during episode of severe sepsis/septic shock will be presented until ICU discharge (for a maximum of 7 days).
Time Frame: Baseline and Days 1-7
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
mL
  Baseline: number analyzed (Participants) | 265 | 187 | 177 | 194 | 558
  Baseline | 3715.19 (2191.23) | 4043.77 (2650.73) | 4250.88 (2943.81) | 3874.96 (2499.80) | 4050.78 (2696.92)
  Day 1: number analyzed (Participants) | 265 | 191 | 177 | 194 | 562
  Day 1 | 2513.84 (2649.60) | 2283.24 (2805.64) | 2083.09 (2684.72) | 1600.21 (2326.52) | 1984.43 (2621.80)
  Day 2: number analyzed (Participants) | 241 | 175 | 160 | 181 | 516
  Day 2 | 3688.96 (4071.55) | 3470.11 (4148.24) | 3114.71 (3588.75) | 2584.89 (3621.66) | 3049.40 (3809.45)
  Day 3: number analyzed (Participants) | 214 | 148 | 147 | 157 | 452
  Day 3 | 4179.02 (5054.24) | 4020.24 (4939.49) | 3684.97 (4584.27) | 3212.04 (4932.67) | 3630.48 (4825.32)
  Day 4: number analyzed (Participants) | 201 | 130 | 130 | 139 | 399
  Day 4 | 4347.58 (6027.04) | 4094.19 (5122.49) | 4633.22 (5855.47) | 3880.32 (5643.93) | 4195.31 (5546.47)
  Day 5: number analyzed (Participants) | 173 | 105 | 114 | 124 | 343
  Day 5 | 4600.67 (6723.02) | 4307.39 (5636.37) | 5126.22 (6910.78) | 4079.52 (6367.01) | 4497.16 (6342.44)
  Day 6: number analyzed (Participants) | 154 | 88 | 92 | 109 | 289
  Day 6 | 4750.10 (7322.08) | 4312.81 (6564.90) | 5263.21 (7595.18) | 4224.47 (7163.95) | 4582.04 (7121.18)
  Day 7: number analyzed (Participants) | 139 | 84 | 87 | 97 | 268
  Day 7 | 4978.66 (7803.61) | 4418.66 (7263.42) | 5628.59 (8471.78) | 4425.98 (7977.33) | 4814.08 (7919.51)

17. Secondary Outcome: Daily Urine Output Until ICU Discharge (for a Maximum of 7 Days)
Time Frame: Baseline and Days 1-7
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
mL/h
  Baseline: number analyzed (Participants) | 265 | 187 | 177 | 194 | 558
  Baseline | 73.726 (94.7641) | 72.944 (82.3338) | 74.530 (92.8984) | 83.773 (86.5417) | 77.212 (87.2301)
  Day 1: number analyzed (Participants) | 265 | 191 | 177 | 194 | 562
  Day 1 | 85.277 (70.3224) | 101.270 (80.4142) | 94.290 (70.9804) | 104.049 (75.8876) | 100.031 (75.9501)
  Day 2: number analyzed (Participants) | 241 | 175 | 160 | 181 | 516
  Day 2 | 88.425 (61.2134) | 89.404 (64.9307) | 88.210 (59.6632) | 92.400 (61.8536) | 90.085 (62.1593)
  Day 3: number analyzed (Participants) | 214 | 148 | 147 | 157 | 452
  Day 3 | 104.124 (67.7586) | 104.833 (66.4533) | 85.403 (61.5660) | 97.312 (67.8895) | 95.902 (65.7529)
  Day 4: number analyzed (Participants) | 201 | 130 | 130 | 139 | 399
  Day 4 | 110.078 (73.3563) | 103.459 (69.8165) | 92.311 (65.0558) | 102.859 (64.2044) | 99.618 (66.3843)
  Day 5: number analyzed (Participants) | 173 | 105 | 114 | 124 | 343
  Day 5 | 116.732 (65.1159) | 110.129 (65.7571) | 100.581 (75.5667) | 117.152 (68.3988) | 109.494 (70.2288)
  Day 6: number analyzed (Participants) | 154 | 88 | 92 | 109 | 289
  Day 6 | 119.087 (65.7102) | 126.512 (83.3418) | 116.799 (79.3092) | 118.269 (72.2910) | 120.311 (77.8633)
  Day 7: number analyzed (Participants) | 139 | 84 | 87 | 97 | 268
  Day 7 | 116.082 (65.9402) | 121.751 (68.1265) | 111.499 (72.8493) | 114.284 (69.5828) | 115.720 (70.0786)

18. Secondary Outcome: Cumulative Urine Output Until ICU Discharge (for a Maximum of 7 Days)
Description: Cumulative urinary output (absolute values) will be presented until ICU discharge (for a maximum of 7 Days).
Time Frame: Baseline and Days 1-7
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
mL
  Baseline: number analyzed (Participants) | 265 | 187 | 177 | 194 | 558
  Baseline | 888.834 (1197.4426) | 898.056 (1020.7890) | 947.843 (1264.9054) | 1017.646 (1076.2691) | 955.426 (1121.3215)
  Day 1: number analyzed (Participants) | 265 | 191 | 177 | 194 | 562
  Day 1 | 2046.658 (1687.7381) | 2430.485 (1929.9400) | 2262.948 (1703.5290) | 2497.173 (1821.3014) | 2400.740 (1822.8019)
  Day 2: number analyzed (Participants) | 241 | 175 | 160 | 181 | 516
  Day 2 | 4343.786 (2909.9212) | 4702.538 (3199.5558) | 4534.714 (2825.1740) | 4814.544 (3091.7350) | 4689.788 (3045.8065)
  Day 3: number analyzed (Participants) | 214 | 148 | 147 | 157 | 452
  Day 3 | 6885.176 (4100.2125) | 7527.805 (4401.3731) | 6587.704 (3849.2099) | 7322.964 (4322.9651) | 7150.914 (4211.3049)
  Day 4: number analyzed (Participants) | 201 | 130 | 130 | 139 | 399
  Day 4 | 9501.722 (5247.5530) | 10239.275 (5486.1180) | 8786.522 (5086.7347) | 9851.841 (5478.3671) | 9630.976 (5377.6356)
  Day 5: number analyzed (Participants) | 173 | 105 | 114 | 124 | 343
  Day 5 | 12600.503 (6293.7322) | 13219.597 (6695.6766) | 11132.418 (6230.4688) | 12795.773 (6400.6821) | 12372.680 (6480.0818)
  Day 6: number analyzed (Participants) | 154 | 88 | 92 | 109 | 289
  Day 6 | 15159.980 (7264.4502) | 16354.712 (7864.2281) | 14522.098 (7391.7707) | 15674.783 (7202.3158) | 15514.875 (7479.2644)
  Day 7: number analyzed (Participants) | 139 | 84 | 87 | 97 | 268
  Day 7 | 17817.979 (8226.0238) | 19269.682 (9081.2013) | 17034.774 (8635.0531) | 18380.119 (8479.7547) | 18222.202 (8736.1728)

19. Secondary Outcome: Utility, Based on the EuroQol Group's 5-dimension 5-level (EQ-5D-5L) Questionnaire, up to Day 180
Description: The EuroQoL-5-Dimensions (EQ-5D™) was used to assess the overall health of each subject. EQ-5D™ is a standardised instrument for use as a measure of health outcome. The first part of the instrument includes 5 dimensions where the subject indicates which of the given statements best describes the health state on the day of questionnaire completion. The second part contains a visual analogue scale (VAS) where the subject indicates how good or bad his or her own health is on the day of questionnaire completion.
  EQ-5D-5L will be analyzed by the index value (Range: 0-1; 0=dead state, 1=full health state), the overall quality-adjusted life year (QALY), and the VAS score (Range: 0-100; 0=worst health state, 100=best health state). The EQ-5D-5L was completed at baseline and at the scheduled follow-up days (i.e. Day 30, Day 60, Day 90, and Day 180).
  Data for EQ VAS score and EQ-5D-5L index score are reported in this endpoint.
Time Frame: Baseline and Days 30, 60, 90 and 180
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
score on a scale
  EQ VAS score (Baseline): number analyzed (Participants) | 166 | 109 | 108 | 129 | 346
  EQ VAS score (Baseline) | 69.2 (21.13) | 69.9 (21.69) | 67.0 (21.60) | 67.4 (22.83) | 68.1 (22.07)
  EQ VAS score (Day 30): number analyzed (Participants) | 130 | 90 | 77 | 88 | 255
  EQ VAS score (Day 30) | 59.4 (21.21) | 54.7 (21.12) | 53.8 (19.63) | 53.9 (23.99) | 54.2 (21.65)
  EQ VAS score (Day 60): number analyzed (Participants) | 132 | 92 | 82 | 87 | 261
  EQ VAS score (Day 60) | 64.5 (20.58) | 62.6 (20.92) | 62.6 (18.94) | 63.8 (20.30) | 63.0 (20.04)
  EQ VAS score (Day 90): number analyzed (Participants) | 130 | 87 | 80 | 87 | 254
  EQ VAS score (Day 90) | 68.2 (19.61) | 65.9 (20.70) | 67.0 (17.50) | 68.1 (18.63) | 67.0 (18.98)
  EQ VAS score (Day 180): number analyzed (Participants) | 129 | 88 | 85 | 86 | 259
  EQ VAS score (Day 180) | 72.6 (20.07) | 71.2 (18.55) | 67.4 (21.39) | 69.7 (20.29) | 69.5 (20.08)
  EQ-5D-5L index score (Baseline): number analyzed (Participants) | 168 | 110 | 109 | 132 | 351
  EQ-5D-5L index score (Baseline) | 0.7305 (0.25098) | 0.7648 (0.22393) | 0.7576 (0.23070) | 0.7380 (0.22152) | 0.7525 (0.22481)
  EQ-5D-5L index score (Day 30): number analyzed (Participants) | 130 | 92 | 80 | 91 | 263
  EQ-5D-5L index score (Day 30) | 0.5706 (0.29463) | 0.5600 (0.27848) | 0.5089 (0.29004) | 0.5283 (0.33580) | 0.5335 (0.30245)
  EQ-5D-5L index score (Day 60): number analyzed (Participants) | 133 | 94 | 83 | 89 | 266
  EQ-5D-5L index score (Day 60) | 0.6707 (0.26160) | 0.6788 (0.22544) | 0.6719 (0.21777) | 0.6746 (0.25391) | 0.6753 (0.23222)
  EQ-5D-5L index score (Day 90): number analyzed (Participants) | 131 | 88 | 81 | 89 | 258
  EQ-5D-5L index score (Day 90) | 0.7207 (0.22523) | 0.7018 (0.26544) | 0.7290 (0.21608) | 0.6810 (0.24960) | 0.7032 (0.24515)
  EQ-5D-5L index score (Day 180): number analyzed (Participants) | 130 | 89 | 88 | 87 | 264
  EQ-5D-5L index score (Day 180) | 0.7627 (0.22170) | 0.7572 (0.19803) | 0.7409 (0.19813) | 0.7435 (0.23729) | 0.7472 (0.21112)

20. Secondary Outcome: Utility, Based on the EuroQol Group's 5-dimension 5-level (EQ-5D-5L) Questionnaire, up to Day 180
Description: The EQ-5D™ was used to assess the overall health of each subject. EQ-5D™ is a standardised instrument for use as a measure of health outcome. The first part of the instrument includes 5 dimensions where the subject indicates which of the given statements best describes the health state on the day of questionnaire completion. The second part contains a VAS where the subject indicates how good or bad his or her own health is on the day of questionnaire completion.
  EQ-5D-5L will be analyzed by the index value (Range: 0-1; 0=dead state, 1=full health state), the overall QALY, and the VAS score (Range: 0-100; 0=worst health state, 100=best health state). The EQ-5D-5L was completed at baseline and at the scheduled follow-up days (i.e. Day 30, Day 60, Day 90, and Day 180).
  Data for EQ-5D-5L QALY is reported in this endpoint.
Time Frame: Days 30, 60, 90 and 180
Population: The FAS comprised of all subjects who were enrolled (i.e. randomized [as planned]) and dosed.
Measure: Mean (Standard Deviation); unit: Quality-adjusted life-year
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
Number analyzed (Participants) | 266 | 191 | 177 | 194 | 562
Quality-adjusted life-year
  EQ-5D-5L QALY (Day 30): number analyzed (Participants) | 125 | 86 | 74 | 86 | 246
  EQ-5D-5L QALY (Day 30) | 0.036 (0.0558) | 0.039 (0.0448) | 0.033 (0.0388) | 0.030 (0.0501) | 0.034 (0.0451)
  EQ-5D-5L QALY (Day 60): number analyzed (Participants) | 126 | 84 | 75 | 82 | 241
  EQ-5D-5L QALY (Day 60) | 0.088 (0.0683) | 0.093 (0.0588) | 0.085 (0.0548) | 0.084 (0.0643) | 0.087 (0.0595)
  EQ-5D-5L QALY (Day 90): number analyzed (Participants) | 123 | 80 | 74 | 82 | 236
  EQ-5D-5L QALY (Day 90) | 0.144 (0.0819) | 0.146 (0.0725) | 0.145 (0.0670) | 0.139 (0.0760) | 0.143 (0.0718)
  EQ-5D-5L QALY (Day 180): number analyzed (Participants) | 120 | 80 | 80 | 81 | 241
  EQ-5D-5L QALY (Day 180) | 0.330 (0.1174) | 0.338 (0.1239) | 0.329 (0.1011) | 0.319 (0.1155) | 0.328 (0.1137)

ADVERSE EVENTS:
Time Frame: All-cause mortality, defined as the percentage of subjects that have died regardless of cause, was recorded up to Day 180. Treatment-emergent adverse events (TEAEs) were collected during the treatment period, i.e., TEAEs occurring after IMP infusion to within 12 hours after the IMP infusion was stopped.
Description: All treated subjects were included in the safety analysis set and were analyzed according to the actual treatment received.
Arm/Group | Placebo | Selepressin 2.5 ng/kg/Min | Selepressin 3.75 ng/kg/Min | Selepressin 5.25 ng/kg/Min | Selepressin Pooled
All-Cause Mortality (participants affected / at risk) | 116/266 | 80/191 | 76/177 | 85/194 | 241/562
Serious Adverse Events (participants affected / at risk) | 85/266 | 57/191 | 65/177 | 57/194 | 179/562
Other Adverse Events (participants affected / at risk) | 94/266 | 54/191 | 63/177 | 60/194 | 177/562
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=266) | Selepressin 2.5 ng/kg/Min (N=191) | Selepressin 3.75 ng/kg/Min (N=177) | Selepressin 5.25 ng/kg/Min (N=194) | Selepressin Pooled (N=562)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic necrosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 5 (7) | 5 (6) | 1 (1) | 11 (14)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial depression (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial stunning (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (3) | 7 (8)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 24 (24) | 10 (10) | 17 (17) | 12 (12) | 39 (39)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 15 (15) | 10 (10) | 12 (12) | 8 (8) | 30 (30)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vasculitis cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 5 (5) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 7 (7)
Shock (Vascular disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Vasoconstriction (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=266) | Selepressin 2.5 ng/kg/Min (N=191) | Selepressin 3.75 ng/kg/Min (N=177) | Selepressin 5.25 ng/kg/Min (N=194) | Selepressin Pooled (N=562)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (13) | 9 (9) | 10 (10) | 11 (11) | 30 (30)
Anaemia (Blood and lymphatic system disorders) | 24 (25) | 12 (13) | 6 (6) | 7 (7) | 25 (26)
Atrial fibrillation (Cardiac disorders) | 30 (43) | 22 (23) | 24 (27) | 22 (29) | 68 (79)
Expired product administered (Injury, poisoning and procedural complications) | 50 (94) | 26 (48) | 29 (47) | 31 (62) | 86 (157)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 9 (9) | 4 (4) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT02508649/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT02508649/SAP_001.pdf